CLINICAL TRIAL: NCT06910514
Title: Multicenter, Randomized, Double-Blind Clinical Trial on the Efficacy and Safety of a Solution for Endoscopic Mucosal Resection of Colonic Lesions
Brief Title: Efficacy and Safety of a Solution for Endoscopic Mucosal Resection of Colonic Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nakafarma S.L. (Industry)
Collaborators: Hospital Torrecárdenas, Almería, Spain (Unknown); Hospital Poniente, El Ejido, Almería, Spain (Unknown); Hospital Virgen del Rocío, Seville, Spain (Unknown); Hospital de Baza, Granada, Spain (Unknown); Hospital Virgen de Valme, Seville, Spain (Unknown); Quirónsalud, Málaga, Spain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEMI-2019-01
Record Dates: First submitted 2025-03-07; First posted 2025-04-04 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Endoscopic Mucosal Resection; Colonic Neoplasms; Therapeutic Irrigation; Treatment Outcome
Keywords: DEMIREX
MeSH Terms: conditions — Colonic Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Double-Blind Clinical Trial with a 4:1 Allocation on the Efficacy and Safety of a Solution for Endoscopic Mucosal Resection of Colonic Lesions
Who Masked: Participant, Investigator
Masking Description: This study is a double-blind, randomized clinical trial, meaning that participants and investigators are unaware of the treatment allocation. The investigational solution and the comparator (placebo or treatment) are identical in appearance, volume, and administration method to ensure blinding. Unblinding will only occur in cases of medical necessity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline solution 0.9% (Placebo Comparator): This arm of the study serves as the placebo comparator, where participants will receive a sterile saline solution administered under the same conditions as the experimental treatment. The saline solution does not contain the active ingredient being studied and will be used to evaluate the efficacy and safety of the experimental treatment in comparison to the control group.
  Interventions: Combination Product: Saline solution 0.9%
- DEMIREX (Experimental): This arm of the study serves as the experimental treatment group, where participants will receive a study solution administered under conditions intended to facilitate endoscopic mucosal resection of colonic lesions. This experimental arm aims to evaluate the efficacy and safety of this novel solution (Demirex) for the endoscopic resection of mucosal lesions in the colon with a diameter of ≥2 cm
  Interventions: Combination Product: Mucopolysaccharide saline solution 0.9%

INTERVENTIONS:
Combination Product: Mucopolysaccharide saline solution 0.9% — Injectable solution designed for submucosal elevation in endoscopic mucosal resection. Administered via submucosal injection prior to polyp resection, adding 1% indigo carmine before administration.
  Arms: DEMIREX
Combination Product: Saline solution 0.9% — Control injectable solution composed of saline 0.9 %. Administered via submucosal injection prior to polyp resection, adding 1% indigo carmine before administration.
  Arms: Saline solution 0.9%

SUMMARY:
The objetive of this clinical trial is to evaluate the efficacy and safety of a solution for endoscopic mucosal resection of colonic lesions in patients undergoing endoscopic resection procedures.

The main questions it aims to answer are:

Does the investigational solution improve the efficacy of endoscopic mucosal resection compared to standard practice? Is the investigational solution safe for use in colonic lesion resection procedures?

Researchers will compare the investigational solution (Demirex) to a standard or placebo solution to see if it improves procedural outcomes and safety profiles.

Participants will undergo endoscopic mucosal resection using either the investigational solution or the comparator, and will be monitored for procedural success, safety, and any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any sex, >18 years old, diagnosed with sessile or flat polyps, with a diameter greater than or equal to 2 cm, in the intestinal submucosa by the Endoscopy Unit.
* The subject has understood and signed an informed consent form (ICF) approved by a Research Ethics Committee (REC) before any study evaluation and commits to completing the study as defined in the protocol.
* Not undergoing active treatment with antiplatelet or anticoagulant drugs.
* After signing the informed consent, patients are scheduled for lesion resection within <3 months from their diagnosis.

Exclusion Criteria:

* Patients with documented allergy to any of the components of the mucosectomy solution or drugs used in sedation.
* Pregnant women.
* Patients on contraceptive treatment or post-menopausal.
* Hematological disorders with uncorrected coagulation abnormalities, with an INR >= 1.5, or patients undergoing active treatment with antiplatelet or anticoagulant drugs.
* Patients with intestinal perforation or obstruction, toxic megacolon, diverticulitis, or inflammatory bowel disease.
* Patients with previous partial resection or pending resection.
* Patients with lesions classified as Paris type III and/or invasive intestinal carcinoma and/or metastases. Patients with previous treatment of the lesion (radiotherapy, endoscopic, surgical, chemotherapy).
* Patients included in another study during the previous month.
* Conditions that, in the medical judgment, contraindicate polyp removal.
* Absence of a signed informed consent, non-acceptance, or contraindication of surgical or anesthetic techniques (Patients with ASA status: High anesthetic risk (ASA score > 3)) and difficulty in the patient's understanding of the conditions of the endoscopic procedure.
* Endoscopic appearance of invasive malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Persistence of the compound in the submucosa | From administration up to 120 minutes post-injection
  Duration for which the injected compound remains visible in the submucosa, assessed through clinical observation and imaging techniques.

SECONDARY OUTCOMES:
Effective duration of the wheal | Every 5 minutes up to 120 minutes post-injection
  Time in minutes during which the wheal remains visible and measurable after the compound injection, assessed using a digital caliper.
Local adverse reactions | Up to 6 months post-injection
  Number of participants experiencing local adverse reactions, evaluated through clinical inspection and classified according to the CTCAE v4.0 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Morales Molina, PhD in Pharmacy, Study Director — Pharmacy Department, Torrecárdenas Hospital, 04009 Almería, Spain; Jose Antonio Morales Molina, PhD in Pharmacy, Principal Investigator — Pharmacy Department, Torrecárdenas Hospital, 04009 Almería, Spain; Sergio Ángel Requejo, Study Chair — NAKAFARMA SL
Locations (1):
- Hospital Universitario Torrecárdenas, Almería, Almería, Spain